CLINICAL TRIAL: NCT06099470
Title: Investigation of the Effects of Synchronized and Non-synchronized Telerehabilitation Programs in the Management of Chronic Non-specific Low Back Pain.
Brief Title: Investigation of the Effects of Telerehabilitation Groups for Chronic Non-specific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yeditepe2023
Record Dates: First submitted 2023-09-19; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Chronic Non-specific Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real-time synchronized telerehabilitation program (STP). (Experimental): Subjects in this group will have face to face real-time video tele-habilitation sessions twice a week using Zoom
  Interventions: Other: Real-time synchronized telerehabilitation program (STP).
- Pre-recording non-synchronized telerehabilitation program (NSTP) (Experimental): Subjects in this group will receive their therapeutic exercises through instructional videos sent via Email or WhatsAPP.
  Interventions: Other: Pre-recording non-synchronized telerehabilitation program (NSTP)
- Home non-supervised control group (HCG) (Other): Minimum intervention which is a PDF file containing the same exercises with no follow ups.
  Interventions: Other: Home non-supervised control group (HCG)

INTERVENTIONS:
Other: Real-time synchronized telerehabilitation program (STP). — patient education, core stabilization exercises, strengthening exercises, stretching exercises
  Arms: Real-time synchronized telerehabilitation program (STP).
Other: Pre-recording non-synchronized telerehabilitation program (NSTP) — Pre-recording non-synchronized telerehabilitation program (NSTP)
  Arms: Pre-recording non-synchronized telerehabilitation program (NSTP)
Other: Home non-supervised control group (HCG) — Home non-supervised control group (HCG)
  Arms: Home non-supervised control group (HCG)

SUMMARY:
The goal of this study is to investigate the efficacy of different internet based delivery methods for patients with chronic non-specific low back pain.

The parameters we want to study is pain, disability, fear of movement, and quality of life.

DETAILED DESCRIPTION:
This study is a randomized control trial with two intervention groups and one control group with total sample size of 72:

1. Real-time synchronized telerehabilitation program (STP). (n=24)
2. Pre-recording non-synchronized telerehabilitation program (NSTP). (n=24)
3. Home non-supervised control group (HCG). (n=24)

Sample Size Calculation:

An adequate sample size was calculated using G*power 3.1.9.7. Statistical test fixed effects one-way ANOVA, the probability for alpha error (α) at 0.05, large effect size f = 0.4, power = 0.8, and three groups. A total of 66 subjects was calculated as the minimum required sample size. In addition, based on previous studies a dropout rate was set at 10%. Hence, the total sample size was increased to 72. Therefore, each group will have 24 subjects (n=24).

Method:

Intervention:

The three groups received a video conference education session. The content of the session was anatomy and physiology of the musculoskeletal structure, and kinesiology of the lumbar region. In addition, they were educated about the principles of pain, possible causes for the CNLBP, and how to manage CNLBP (correct posture and life modifications).

Subjects in the STP and NSTP received the same exercises based on core stabilization and stretching but with different method.

1. STP group will benefit from individual exercise session through real-time video calls, where the therapist demonstrates the exercises, and monitor the patient throughout the session.
2. NSTP group will benefit from thoroughly instructional videos that describe every step of each exercise and will be followed up weekly through a video call to monitor compliance and answer questions.
3. HCG group will receive a PDF file that includes the same exercises with written instructions. However, no further interventions nor follow-ups will be available for the HCG.

Protocol:

The exercise protocol (table1) will be as follow with total duration of 44 minutes:

Warm-up (5 minutes): Head tilt, head rotation, shoulder circles, chest stretch, side bend, hip circles, torso twist, forward bend, Cat-cow.

Stabilization exercises (25 minutes):

1. Level one: Tabletop with single knee and hip flexion. 4-point kneeling with single leg stretch. Bridge. One leg stretch. Straight leg side lifts. Sit-ups with lumbar region fixed on the floor.
2. Level two: Tabletop with step knee and hip flexion. 4-point kneeling with single-leg rise. Bridge with leg stretch. One leg stretch with knee extension. Straight leg side lifts with contralateral adduction. Sit-ups reach wrists to the knees.
3. Level three: Tabletop with double knee and hip flexion. 4-point kneeling with contralateral arm and leg raise. Bridge with leg stretch and hold. One leg stretch hold and alternate knee extension. Straight leg side lifts adduct and hold. Sit-ups arms crossed over the chest.

   * 10 repetitions, 10 seconds rest intervals, 3 sets. Cooldown and stretching exercises (14 minutes): quadriceps stretch, kneeling hip flexor stretch, sitting adductor stretch, seated hip and ITB stretch, gluteal stretch (in prone position), piriformis stretch, hamstring-gastrocnemius stretch with a band, abdominal stretch, bend forward stretch.

     30 seconds hold for each exercise, 3 cycles.

ELIGIBILITY:
Inclusion criteria

* Persisting low back pain for the past 3 months.
* VAS score of at least 4.
* Age between 18 and 65.
* Ability to perform exercises.
* Internet access.

Exclusion criteria

* Pregnancy.
* History of spinal surgery.
* History of spinal injury.
* Misalignment or specific condition in the lumbar region.
* Inflammatory joint diseases.
* Any neurological symptoms.
* Diagnosed osteoporosis.
* Spondylosis.
* Radiculopathy in the lumbar region.
* Having a current inflammation in the trunk, lumbar or pelvic region.
* Receiving physical therapy or other conventional therapy for LBP in the past 6 months.
* Regular practice for Pilates or other specific exercise programs in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 12 weeks
  is a visual scale with various types to measure the intensity of the pain where 0 is considered no pain and 10 is unbearable pain. VAS can be just a 100mm horizontal line where patients can put a mark anywhere on the line, or graphics indicating the severity of pain. Also, it can be numerical line from 0 to 10 which we intend to use in this thesis.

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire | 12 weeks
  A sensitive and reliable evaluation tool, to measure disability in patients with chronic non-specific low back pain. It contains a 24-item scale with a total score ranging from 0 (no disability) to 24 (high disability). The questionnaire was prepared in the questionnaire was delivered electronically as checkboxes question on the prepared assessment google forms.
  Patients were asked to only choose the sentences that describes how they feel today and skip the sentences that does not.
Oswestry Disability Index | 12 weeks
  Is a gold standard, valid questionnaire, which assesses disability in ten distinct parts: pain intensity, patient personal care, lifting, walking, sitting, standing, sleeping, social life, sex life and travelling. Each statement is scored from 0 to 5 with higher scores demonstrating more disability. The questionnaire was prepared and delivered electronically as ten multiple choice questions on the prepared assessment google forms.
  Patients were asked to choose the part that most closely describes how they feel today.
Tampa Scale for Kinesiophobia | 12 weeks
  Tampa Scale for Kinesiophobia (TSK) was used. Which is a reliable 17-item scale to measure fear of movement and injury in patients with CNLBP. Each item ranges from 1 to 4 points, with 1 point for "total disagree," to 4 points for "total agree". The total score of the scale ranges from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia
SF-12 Health Questionnaire | 12 weeks
  SF-12 Health Questionnaire was used. Which is a questionnaire that measures the quality of life, by assessing the impact of health on everyday activities. It uses the same eight domains as the SF-36: limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems, limitations in usual role activities because of physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities because of emotional problems, vitality (energy and fatigue), general health perceptions. The questionnaire was prepared and delivered electronically as 12 multiple choice questions on the prepared assessment google forms.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe ÇİL, Dr, Study Chair — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Sipaviciene S, Kliziene I. Effect of different exercise programs on non-specific chronic low back pain and disability in people who perform sedentary work. Clin Biomech (Bristol). 2020 Mar;73:17-27. doi: 10.1016/j.clinbiomech.2019.12.028. Epub 2020 Jan 3. PMID 31923778
- [Background] In TS, Jung JH, Jung KS, Cho HY. Effects of the Multidimensional Treatment on Pain, Disability, and Sitting Posture in Patients with Low Back Pain: A Randomized Controlled Trial. Pain Res Manag. 2021 Jun 30;2021:5581491. doi: 10.1155/2021/5581491. eCollection 2021. PMID 34306274
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Narouei S, Barati AH, Akuzawa H, Talebian S, Ghiasi F, Akbari A, Alizadeh MH. Effects of core stabilization exercises on thickness and activity of trunk and hip muscles in subjects with nonspecific chronic low back pain. J Bodyw Mov Ther. 2020 Oct;24(4):138-146. doi: 10.1016/j.jbmt.2020.06.026. Epub 2020 Jul 30. PMID 33218502
- [Background] Zhang Y, Tang S, Chen G, Liu Y. Chinese massage combined with core stability exercises for nonspecific low back pain: a randomized controlled trial. Complement Ther Med. 2015 Feb;23(1):1-6. doi: 10.1016/j.ctim.2014.12.005. Epub 2015 Jan 3. PMID 25637146
- [Background] Macedo LG, Maher CG, Latimer J, McAuley JH. Motor control exercise for persistent, nonspecific low back pain: a systematic review. Phys Ther. 2009 Jan;89(1):9-25. doi: 10.2522/ptj.20080103. Epub 2008 Dec 4. PMID 19056854
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533
- [Background] Paatelma M, Kilpikoski S, Simonen R, Heinonen A, Alen M, Videman T. Orthopaedic manual therapy, McKenzie method or advice only for low back pain in working adults: a randomized controlled trial with one year follow-up. J Rehabil Med. 2008 Nov;40(10):858-63. doi: 10.2340/16501977-0262. PMID 19242624